CLINICAL TRIAL: NCT01163370
Title: Creatine Supplementation and Bone Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: creatine and bone
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Osteopenia; Osteoporosis
Keywords: creatine supplementation; resistance training; osteopenia; osteoporosis; bone mineral density
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Creatine; Exercise; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- control and exercise (Placebo Comparator): this is trained and receives placebo
  Interventions: Other: exercise training; Other: placebo (dextrose)
- creatine (Experimental): this is non-exercise trained and receives creatine supplementation
  Interventions: Dietary Supplement: creatine supplementation
- exercise and creatine (Experimental): this is exercised trained and receives creatine supplementation
  Interventions: Dietary Supplement: creatine supplementation; Other: exercise training
- placebo (Placebo Comparator): this only receives placebo (dextrose)
  Interventions: Other: placebo (dextrose)

INTERVENTIONS:
Dietary Supplement: creatine supplementation — 20g/d for 7 days followed by 5g/d for 23 weeks
  Arms: creatine; exercise and creatine
Other: exercise training — resistance training twice a week for 24 weeks
  Arms: control and exercise; exercise and creatine
Other: placebo (dextrose) — 20g/d for 7 days followed by 5g/d for 23 weeks
  Arms: control and exercise; placebo

SUMMARY:
Resistance training as well as creatine supplementation may increase bone mass. Therefore, the investigators speculate that resistance training combined with creatine supplementation would promote additive benefits on bone mass in elderly women with osteopenia and osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* osteopenia and osteoporosis
* women older than 60 years old

Exclusion Criteria:

* cardiovascular diseases or muscular disturbances precluding exercise training
* drugs affecting bone metabolism

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
bone mineral density | six months

SECONDARY OUTCOMES:
cognition | six months
physical capacity | six months
  including muscle strength, balance and muscle function

CONTACTS AND LOCATIONS:
Overall Officials: Rosa MR Pereira, PhD, Principal Investigator — University of Sao Paulo; Bruno Gualano, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Medicine - Division of Rheumatology, São Paulo, São Paulo, Brazil